CLINICAL TRIAL: NCT04815187
Title: Repurposed Use of Allergic Rhinitis and Allergic Asthma Drug to Reduce Vertigo and Hearing Loss in Meniere's Disease
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: House Ear Institute (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20203338
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Meniere Disease; Allergic Rhinitis; Vertigo
MeSH Terms: conditions — Meniere Disease; Rhinitis, Allergic; Vertigo | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Montelukast 10 mg (Experimental): Subjects will be instructed to take one pill at night for 90 days
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Subjects will be instructed to take one pill at night for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Each subject will be given a drug diary to record when they took the drug and any symptoms that they are experiencing, and will bring this diary and any unused pills to their next clinic visit before receiving the next 30-day supply. This process will continue for the full 90 days of study involvement, with a final visit 3 months later.
  Arms: Montelukast 10 mg
Drug: Placebo — Each subject will be given a drug diary to record when they took the drug and any symptoms that they are experiencing, and will bring this diary and any unused pills to their next clinic visit before receiving the next 30-day supply. This process will continue for the full 90 days of study involvement, with a final visit 3 months later.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate a previously FDA-approved medication that is known to help with allergy symptoms to see if it can decrease symptoms in patients with Meniere's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Must meet all AAO-HNS 2020 criteria for definite or probable Meniere's Disease
* Must have a skin test positive for allergy
* Is already a candidate for treatment with montelukast for allergic rhinitis/failed first line over-the-counter allergy treatments

Exclusion Criteria:

* Had a previous surgical procedure for treatment of vertigo
* Currently receiving any allergy immunotherapy or taking montelukast or a beta-blocker
* Pregnant or recent pregnancy ((≤ 8 weeks postpartum), or lactation)
* Current hospitalization for any reason
* Any active, acute, or chronic pulmonary disorder other than asthma
* History of intubation for asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients with AAO-HNS Vertigo Control Class A or B | 1 month after treatment initiation
  Percentage of patients in each group with an AAO-HNS Vertigo Control Class A or B result (from daily diary count of number of attacks)
Percentage of Patients with AAO-HNS Vertigo Control Class A or B | 3 months after treatment initiation
  Percentage of patients in each group with an AAO-HNS Vertigo Control Class A or B result (from daily diary count of number of attacks)
Percentage of Patients with AAO-HNS Vertigo Control Class A or B | 6 months after treatment initiation
  Percentage of patients in each group with an AAO-HNS Vertigo Control Class A or B result (from daily diary count of number of attacks)
Difference in Dizziness Between Treatment Arms | 3 months after treatment initiation
  Difference for each group in AAO-HNS dizziness functional disability scale from pre-treatment to 3 months after treatment initiation. A score improvement of 1 point on this 6-point scale will be considered significant improvement.
Percentage of Subjects Experiencing Significant Hearing Fluctuation | 3 months after treatment initiation
  Percentage of subjects in each treatment arm demonstrating clinically significant change in air conduction thresholds at > 2 frequencies at 3 months (> 10 dB change from baseline) or WDS (> 15% change from baseline) compared to the worst audiogram and WDS in the 6 months prior to treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Derebery, MD, Principal Investigator — House Institute Foundation
Locations (2):
- United States (2):
  - House Ear Clinic, Los Angeles, California
  - House Institute Foundation, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No